CLINICAL TRIAL: NCT04760106
Title: The Feasibility of Ultrasound for the Qualitative Assessment of Gastric Content, and Determine the Reliability of This Novel Tool in Gastric Volume Measurements When Performed by Novice Gastric Sonographers
Brief Title: Learning Curves of Gastric Ultrasound for Novel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si 830/2018
Record Dates: First submitted 2021-02-07; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Gastric Ultrasound; Learning Curve; Novel in Gastric Ultrasound
Keywords: Gastric ultrasound; Learning curve; Accuracy; Reliability; Novel in gastric ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: gastric ultrasound — For the qualitative assessment, every participant was scanned once by both examiners. Each scan session lasted no longer than 5 minutes to mitigate the confounding effect of gastric emptying time.
  For the quantitative assessment, the participants were put in a right lateral decubitus position and the antral cross-sectional area (CSA) is measured in the sagittal plane.

SUMMARY:
Various studies have shown that gastric sonography can reliably provide information on both qualitative (nature of content) and quantitative (volume) aspects of gastric content. A recent study has suggested that a minimum of 33 scans is needed to achieve a 95% success rate in the qualitative assessment of gastric ultrasound. However, as the risk and severity of aspiration are also influenced by gastric volume, further study concerning quantitative assessment is warranted.

DETAILED DESCRIPTION:
This study are conducted to affirm the feasibility of ultrasound for the qualitative assessment of gastric content, and determine the reliability of this novel tool in gastric volume measurements when performed by novice gastric sonographers. Two novels in gastric ultrasound learn from online materials, including educational videos and picture library through www.gastricultrasound.org and www.usra.ca. 1-hour lecture with discussion and 1-hour interactive hands-on with expert in gastric ultrasound. Then the novels were tested for the accuracy and reliability of their skills from 50 volunteers gastric ultrasound assessment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 70 years old with an American Society of Anesthesiologist physical status class I to II

Exclusion Criteria:

* BMI > 40 kg/m2; pregnancy; diabetes mellitus; a history of upper gastrointestinal tract disease (including hiatal hernia and gastric tumors); and previous surgical procedures on the esophagus, stomach, or upper abdomen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The accuracy of qualitative ultrasound assessment of gastric content in novel gastric sonographers | 3 months
  Number of volunteers which novel gastric sonographers are correct to identify whether is empty, fluid or solid (percentage)

SECONDARY OUTCOMES:
An interrater reliability of the quantitative ultrasound assessment of the gastric volume | 3 months
  Using the result of cross sectional area from both novel gastric sonographers

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tankul R, Halilamien P, Tangwiwat S, Dejarkom S, Pangthipampai P. Qualitative and quantitative gastric ultrasound assessment in highly skilled regional anesthesiologists. BMC Anesthesiol. 2022 Jan 3;22(1):5. doi: 10.1186/s12871-021-01550-z. PMID 34979932